CLINICAL TRIAL: NCT04260139
Title: Macroscopic Evaluation of Colon Cancer Resection Specimens to Predict Metastatic Lymph Node Yield
Brief Title: Lymph Node Yield in Colon Cancer Resection Specimens
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nadir Adnan Hacım, Dr., Bagcilar Training and Research Hospital
Other Study IDs: Beren Hacım
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Colon Cancer; Lymph Node Metastases
Keywords: ileocolic pedicle; colon cancer; Staging
MeSH Terms: conditions — Colonic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Calculation of metric variables on the colectomy specimens. — Calculation of metric variables on the colectomy specimens including Lengths as mm
  1. Proximal colon,
  2. Ileum in cases with right hemicolectomy only,
  3. Proximal border,
  4. Tumor,
  5. Distal border,
  6. Total specimen,
  7. Vascular pedicle, the longitudinal distance between the nearest bowel wall and the end of ligated major vascular pedicle depending on the tumor's localization, 2. Colonic mesenteric area as mm2.

SUMMARY:
In this study, we aimed to develop a predictive model of lymph node yield in a series of colon cancer resection specimens with detailed anatomic and surgical technique data.

DETAILED DESCRIPTION:
Lymph node yield in colon resection specimens has been associated with the accuracy of staging and cancer outcomes. It has been proposed that the more central the mesenteric vascular ligation, the greater the nodal yield. However, the optimal number of harvested nodes is still a matter of debate. We prospectively evaluated the relation between specimen properties such as lenght, area, tumor location and pedicle length to the number of harvested nodes and rate of node positivity.

ELIGIBILITY:
Inclusion Criteria:

The surgical patients with a histologic diagnosis of colonic neoplasm, Colectomy of any type, including the right hemicolectomy, the left hemicolectomy, the sigmoid resection, segmental colon resection

Exclusion Criteria:

* rectal or rectosigmoid cancer colectomy beyond the inclusion criteria for colectomies patients younger than 18 previous colon resection emergency colon resection familial adenomatous polyposis or ulcerative colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pathology specimens from colon neoplasm resections will be prepared so that the lymph nodes will be separated according to their anatomic relationship to the vascular pedicles and to the tumor. Prior to dissection, the specimen will be measured from all colonic tumor patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Lymph Node Yield in Colon Cancer Resection Specimens | September 2019- November 2020
  Count of lymph node
Lymph Node Yield in Colon Cancer Resection Specimens | September 2019-November 2020
  Involvement of lymph node

CONTACTS AND LOCATIONS:
Locations (1):
- Bagcılar Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No